CLINICAL TRIAL: NCT00287300
Title: A Pilot Randomized Controlled Trial of Azithromycin or Artesunate Added to Sulphadoxine Pyrimethamine as Therapy for Malaria in Pregnancy
Brief Title: Efficacy and Safety of Azithromycin and Artesunate in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03-EPID-153
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2006-02-06 (Estimated); Status verified 2006-01

CONDITIONS: Malaria
Keywords: Malaria; Pregnancy; Efficacy; Azithromycin; Artesunate
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Azithromycin; Artesunate

INTERVENTIONS:
Drug: Sulfadoxine-Pyrimethamine
Drug: Azithromycin
Drug: Artesunate

SUMMARY:
The purpose of this study is to compare the efficacy and safety of three treatment regimens for the prevention of malaria during pregnancy.

DETAILED DESCRIPTION:
Malaria infection during pregnancy poses substantial risk to the mother, her fetus, and the neonate. Prevention of malaria during pregnancy is vital in decreasing maternal and child mortality in Africa. There are data from studies that show that intermittent preventive treatment (IPT) with two doses of sulfadoxine-pyrimethamine (SP) is safe, efficacious, and effective in preventing maternal anemia, placental parasitemia, and LBW. Resistance to SP, however, is increasing rapidly in Africa and there is an urgent need to find alternative effective, safe and affordable drugs for the treatment and prevention of malaria in pregnancy.

The investigators conducted a trial to determine the efficacy and safety of azithromycin and artesunate combined with sulphadoxine-pyrimethamine as treatment against malaria during pregnancy.Pregnant women 14 to 26 weeks gestation with P. falciparum parasitemia on peripheral blood film were randomly assigned into 3 treatment groups and received two doses of:(1) SP (3 tablets) only; (2) SP and azithromycin (1gram/day x 2 days)and (3) SP and artesunate 200mg/day for 3 days). The two doses of the study drug were administered approximately 4 weeks apart. All study drugs were taken under observation.Blood samples were collected on days 1, 2, 3, 7 and 14 after treatment and at any visit when the women presented with symptoms of malaria. The women were also given an insecticide-treated net (ITN) and followed until delivery. Adverse effects were assessed at each scheduled visit, any unscheduled visits during the study, and at delivery. Peripheral and placental blood films and placental biopsies were prepared at delivery. Newborns were weighed, examined, and gestational age was determined.

ELIGIBILITY:
Inclusion Criteria:

* peripheral malaria parasitemia
* signed informed consent
* age 15-49 years
* mother has felt the movements of the foetus (quickening)
* fetal age of at least 14 but not more than 26 completed gestation weeks
* maternal availability for follow-up during the entire period of the study

Exclusion Criteria:

* known maternal tuberculosis, diabetes, kidney disease, or liver disease
* mental disorder that may affect comprehension of the study or success of follow-up
* twin pregnancy
* pregnancy complications evident at enrollment visit (moderate to severe oedema, blood Hb concentration < 7 g / dl, systolic blood pressure (BP) > 160 mmHg or diastolic BP > 100 mmHg)
* prior receipt of azithromycin during current pregnancy
* receipt of any antimalarial within 28 days before enrollment
* known allergy to drugs containing sulfonamides, macrolides or pyrimethamine
* history of anaphylaxis
* history of any serious allergic reaction to any substance, requiring emergency medical care
* history of hepatitis or jaundice
* concurrent participation in any other clinical trial

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 141
Dates: Start 2003-09; Study Completion 2005-08

PRIMARY OUTCOMES:
Parasitological failure rates
Parasite clearance time
Fever clearance times
Incidence rate of adverse events

SECONDARY OUTCOMES:
Prevalence rate of abortions
Prevalence rate of still births
Prevalence rate of peripheral parasitemia at delivery
Prevalence of placental malaria (thick blood film and histology)
Prevalence rate of maternal anemia

CONTACTS AND LOCATIONS:
Overall Officials: Steve R Meshnick, M.D., Ph.D., Principal Investigator — 2. Department of Epidemiology, School of Public Health, University of North Carolina, Chapel Hill NC USA; Stephen J Rogerson, MB BS, Ph.D., Principal Investigator — 3. Department of Medicine, University of Melbourne, Royal Melbourne Hospital, Parkville Victoria Australia; Marjorie Chaponda, MB BS, MPH, Principal Investigator — 1. UNC Malaria Project, Department of Community Health, College of Medicine, University of Malawi
Locations (1):
- Mpemba and Madziabango Health Centers, Blantyre, Malawi

REFERENCES:
- [Derived] Kalilani L, Mofolo I, Chaponda M, Rogerson SJ, Alker AP, Kwiek JJ, Meshnick SR. A randomized controlled pilot trial of azithromycin or artesunate added to sulfadoxine-pyrimethamine as treatment for malaria in pregnant women. PLoS One. 2007 Nov 14;2(11):e1166. doi: 10.1371/journal.pone.0001166. PMID 18000538